CLINICAL TRIAL: NCT05337800
Title: The Effect of Stress Management Program on Clinical Stress of First Year Nursing Students
Brief Title: Stress Management on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Emel Gülnar, assistant professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KirikkaleU12345
Record Dates: First submitted 2022-04-07; First posted 2022-04-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stress; Clinical Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stress management program (Experimental)
  Interventions: Behavioral: stress managment program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: stress managment program — A four-session stress management program will be applied to the experimental group students.
  Arms: stress management program

SUMMARY:
In this study, it was aimed to determine the effect of the stress management program on the clinical stress of first year nursing students. This research will be carried out in a randomized controlled experimental design.

The data of the research; The descriptive characteristics form will be collected using the Perceived Stress Scale for Nursing Students, the Bio-Psycho-Social Response Scale for Nursing Students, and the Stress Coping Behaviors Scale for Nursing Students. students will be assigned as experiment (32) and control (32) by randomization. A four-session stress management program will be applied to the experimental group students. No intervention will be made on the control group.

ELIGIBILITY:
Inclusion Criteria:

The first to enroll in the Nursing Fundamentals course,

Exclusion Criteria:

* Have previously taken nursing fundamentals course

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale for Nursing Students | 15 minute
  It measures the perceived stress of nursing students. It is a Likert type scale and consists of 29 items. Total score; 0 - 116. A high score indicates a higher level of stress.
Bio-Psycho-Social Response Scale for Nursing Students | 20 minute
  It consists of 21 items related to the symptoms related to the physical, psychological and social health of students. It is a Likert type scale and consists of 21 items. Total score; It ranges from 0 to 84. A high score indicates more symptom presence and poor bio-psycho-social status.
Stress Coping Behaviors Scale for Nursing Students | 15 minute
  It measures the stress coping behaviors of students. It consists of 19 items in total. A higher score on a factor indicates that this coping type is used more frequently.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mackenzie CS, Poulin PA, Seidman-Carlson R. A brief mindfulness-based stress reduction intervention for nurses and nurse aides. Appl Nurs Res. 2006 May;19(2):105-9. doi: 10.1016/j.apnr.2005.08.002. PMID 16728295
- [Background] Botha E, Gwin T, Purpora C. The effectiveness of mindfulness based programs in reducing stress experienced by nurses in adult hospital settings: a systematic review of quantitative evidence protocol. JBI Database System Rev Implement Rep. 2015 Oct;13(10):21-9. doi: 10.11124/jbisrir-2015-2380. PMID 26571279
- [Background] Karaca A, Sisman NY. Effects of a Stress Management Training Program With Mindfulness-Based Stress Reduction. J Nurs Educ. 2019 May 1;58(5):273-280. doi: 10.3928/01484834-20190422-05. PMID 31039261